CLINICAL TRIAL: NCT04067739
Title: ICU Readmission in Adult Egyptian Patients Undergoing Living Donor Liver Transplant: Incidence, Causes and Outcomes: A Single Centre Retrospective Observational Study
Brief Title: ICU Readmission in Adult Egyptian Patients Undergoing Living Donor Liver Transplant
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hanaa Mohamed Abdallah ElGendy MD, Assistant Professor, Ain Shams University
Other Study IDs: IRB//0006379
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: ICU Readmission

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Readmission group: Readmission is defined as ICU readmission within ≤ 3 months of initial ICU discharge
  Interventions: Other: non interventional study
- Non readmitted group: Non readmission is defined as no need for ICU readmission within ≤ 3 months of initial ICU discharge
  Interventions: Other: non interventional study

INTERVENTIONS:
Other: non interventional study — non interventional study

SUMMARY:
Liver transplantation is the only definitive treatment for end stage liver disease. Being a major abdominal surgery, may have postoperative complications that require readmission, which may be serious and life threatening. In general, patients who required ICU readmission showed higher morbidity, mortality and prolonged hospital stay compared to those who did not require readmission. We will conduct this retrospective observational study to identify incidence, causes and outcomes of ICU readmission after LDLT

DETAILED DESCRIPTION:
* This retrospective observational study will be conducted in Ain Shams University Specialized Hospital on 335 adult (age ≥18 years) Egyptian patients undergoing living donor liver transplant (LDLT) between 2008 to 2018. Patients' demographic data, preoperative variables, intraoperative variables, postoperative stay and complications, causes for ICU readmission, and outcomes after ICU readmission will be studied. Intraoperatively, Both standard anesthetic and piggyback LT for hepatic transplantation were performed by the same anesthesia and surgical team . Intraoperative patients were monitored with ECG, invasive arterial blood pressure (left radial artery), noninvasive blood pressure, continuous central venous pressure (CVP), body temperature, oxygen saturation (SaO2), capnometry (EtCO2) and urine output (mL). Intraoperative hemodynamics (MAP and HR), graft weight to recipient weight ratio (GWRWR), blood products transfused and intraoperative adverse events were recorded. At the end of surgery patients were transferred to the ICU where they were monitored and received the standard protocol for postoperative management after liver transplantation.
* The postoperative immunosuppressive protocols includes calcinurine inhibitors( FK or cyclosporine), and steroids with or without mycophynolate. Piperacillin/ tazobactam was used as early prophylaxis for bacterial infections and metronidazole as prophylaxis for anaerobic infection. Patients with an uncomplicated postoperative course and good liver function will be transferred from the ICU within 3 - 5 days to a designated transplantation inpatient unit where they will be closely followed up by surgical and medical team, as well as by pharmacists, nutritionists, and physical therapists.

ELIGIBILITY:
Inclusion Criteria:

* Adult Egyptian Patients >18 years

Exclusion Criteria:

* Patient refusal.
* Patients who were not discharged after LDLT due to death.
* Patients who underwent re-transplantation before discharge from the ICU after the first liver transplant.
* Pregnancy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients' demographic data, preoperative variables, intraoperative variables, postoperative stay and complications, causes for ICU readmission, and outcomes after ICU readmission will be studied.Intraoperatively patients were monitored. Intraoperative adverse events were recorded. At the end of surgery patients were transferred to the ICU.
  - The postoperative immunosuppressive protocols includes calcinurine inhibitors( FK or cyclosporine), and steroids with or without mycophynolate. Piperacillin/ tazobactam was used as early prophylaxis for bacterial infections and metronidazole as prophylaxis for anaerobic infection. Patients with an uncomplicated postoperative course and good liver function will be transferred from the ICU within 3 - 5 days to a designated transplantation inpatient unit.
Sampling Method: Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
ICU readmission within ≤ 3 months of initial ICU discharge | within 3 months
  Incidence, causes and outcomes of ICU readmission within ≤ 3 months of initial ICU discharge

SECONDARY OUTCOMES:
one year survival | Within 3 months
  comparison between one year survival in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Hanaa El Gendy, Cairo, Ain Shams University Specialized Hospital, Egypt

IPD SHARING:
Plan to Share IPD: No